CLINICAL TRIAL: NCT00550420
Title: An Open-label Extension to Study AVA105640, to Assess the Long-term Safety and Efficacy of Rosiglitazone (Extended Release Tablets) on Cognition in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: Study Of Rosiglitazone XR In Subjects With Mild-to-Moderate Alzheimers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on preliminary parent study results
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA102677
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease
Keywords: open-label extension; tolerability; Alzheimer's disease; Rosiglitazone extended-release (XR); safety; cognition; BRL-049653
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- Arm 1 (Experimental): Rosiglitazone XR
  Interventions: Drug: Rosiglitazone XR

INTERVENTIONS:
Drug: Rosiglitazone XR — experimental drug

SUMMARY:
This is a Phase III, multicenter, open-label extension, single-group study in male and female outpatients with mild-to-moderate Alzheimer's disease (AD) who have completed AVA105640. All subjects will receive rosiglitazone extended-release (RSG XR) 4mg once daily for the first 4 weeks of the study followed by 8mg RSG XR. Subject participation will last until one of 5 conditions applies. After a 52-week open-label treatment phase, subjects will attend a final Follow-Up Visit 6 weeks after the end of treatment. The primary objective of this study is to evaluate the long-term safety and tolerability of RSG XR in subjects with mild-to-moderate AD who have completed AVA105640. The secondary objective of this study is to explore further the long-term efficacy of RSG XR in terms of cognitive function and overall clinical response as a function of apolipoprotein E (APOE) e4 allele status

ELIGIBILITY:
Inclusion criteria:

* Male or female subject who has successfully completed Visit 8 of AVA105640 without safety/tolerability issues, where in the opinion of the subject /carer and of the investigator, it would be beneficial to receive RSG XR
* Female subjects able to bear children must agree to use an adequate method of contraception for the duration of the study for details of highly effective methods to avoid pregnancy). Female subjects who are pre-menopausal or who have been post-menopausal for <1 year must undertake pregnancy testing (urine test) £7 days before Visit 1, which must be negative
* Subject is willing to participate in the extension study and has provided full written informed consent prior to the performance of any protocol-specified procedure; or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative (where this is in accordance with local laws, regulations and ethics committee policy)
* Subject lives with (or has substantial periods of contact with) a regular caregiver who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status
* Subject has the ability to comply with procedures for cognitive and other testing
* Caregiver has provided full written informed consent on his or her own behalf prior to the performance of any protocol-specified procedure
* Subjects considered for enrollment must have a QTc (either QTc B (Bazett's correction) or QTc F (Fridericia's correction)) <450msec at Visit 1, with the exception of subjects with bundle branch block (for whom either QTc B or QTc F must be <480msec)
* In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category
* Post-menopause [Becker, 2001]: Menopause is the age associated with complete cessation of menstrual cycles, menses, and implies the loss of reproductive potential by ovarian failure. This typically occurs around age 50, although it may occur earlier. A practical definition accepts menopause after one year without menses with an appropriate clinical profile, e.g., age appropriate, >45 years, in the absence of hormone replacement therapy. In questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory (these levels are suggested guidelines and may need to be adjusted for specific laboratories/assays
* Females, who are on hormone replacement therapy (HRT), and whose menopausal status is in doubt, will be required to use a highly effective method to avoid pregnancy, as outlined in the protocol, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw as detailed in the preceding paragraph; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a highly effective method to avoid pregnancy
* A non-cohabiting caregiver must spend sufficient time with the subject so that, in the opinion of the Investigator, the caregiver can reliably assess cognitive function, activities and behaviour, and report on the subject's compliance and health. As caregiver time spent with a potential subject is anticipated to be highly variable across countries and cultures, GSK will consider a variety of different measures by which this stipulation may be met, and GSK should be consulted if adequacy of a caregiver situation is in doubt. However, as guidance, the ability for a caregiver to meet his/her expected responsibilities for this study would normally be possible when the caregiver spends no less than 10 hours per week with the subject, divided over multiple days
* For the purposes of these criteria, QTc B is defined as (QT interval [msec]) / (square root of RR interval [seconds]); and QTc F is defined as (QT interval [msec]) / (cube root of RR interval [seconds])

Exclusion criteria:

* Subject had a serious adverse experience or clinically significant laboratory abnormality during AVA105640, which in the opinion of the investigator could have been attributable to study medication, and which is ongoing at Visit 1
* The subject is felt by the investigator to be unsuitable (on the basis of health, compliance, caregiver availability, or for any other reason) for inclusion in the study
* The subject experienced a significant cardiovascular event during AVA105640 (e.g. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina] or significant arrhythmia), unless a thorough cardiovascular evaluation has been performed which confirms that the subject does not have congestive heart failure, and is clinically stable
* Clinical/investigational evidence of congestive heart failure defined by the New York Heart Association (NYHA) criteria (Class I to IV cardiac status) at the time of Visit 1
* Clinically significant peripheral oedema at the time of Visit 1
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase values >2.5 times the upper limit of normal (ULN), total bilirubin values >1.5 times the ULN, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C)
* Subject is an immediate family member or employee of the participating Investigator, of any of the participating site staff, or of GSK
* In France, a subject is neither affiliated with nor a beneficiary of a social security category
* In France, a subject has participated in any study using an investigational drug during the previous 30 days (except for participation in AVA105640)

Ages: 51 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2007-10-01 (Actual); Primary Completion 2009-02-12 (Actual); Study Completion 2009-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (56):
- United States (9):
  - GSK Investigational Site, Palo Alto, California
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Nashville, Tennessee
- Austria (2):
  - GSK Investigational Site, Graz-Eggenberg
  - GSK Investigational Site, Hall in Tirol
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- China (4):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- GSK Investigational Site, Zagreb, Croatia
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (18):
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Günzburg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Baesweiler, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Jülich, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- Hungary (2):
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
- Mexico (3):
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, México
- GSK Investigational Site, Auckland, New Zealand
- GSK Investigational Site, Lima, Peru
- GSK Investigational Site, Pasig, Philippines
- GSK Investigational Site, San Juan, Puerto Rico
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Korea (2):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- GSK Investigational Site, West of Scotland Science Park, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gold M, Alderton C, Zvartau-Hind M, Egginton S, Saunders AM, Irizarry M, Craft S, Landreth G, Linnamagi U, Sawchak S. Rosiglitazone monotherapy in mild-to-moderate Alzheimer's disease: results from a randomized, double-blind, placebo-controlled phase III study. Dement Geriatr Cogn Disord. 2010;30(2):131-46. doi: 10.1159/000318845. Epub 2010 Aug 21. PMID 20733306
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVA102677 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 331 participants who had completed the double-blind treatment phase in AVA105640 were enrolled. Only 26 participants completed the study as it was early terminated, 206 participants were still enrolled at the time of study termination while 97 participants withdrew prematurely. The study completion status of 2 participants was missing.
Pre-assignment Details: The enrolled participants had successfully completed Visit 8 of AVA105640 without safety/tolerability issues. For safety endpoints, 'baseline' referred to the current study baseline assessment, (AVA102677 Visit 1). For efficacy endpoints, the term 'baseline' referred to the baseline assessment of the parent study (AVA105640), Visit 3.
Groups:
- RSG XR 8 mg: Participants received rosiglitazone extended-release (RSG XR) 4 milligram (mg) tablet once daily, orally for the first 4 weeks of the study followed by RSG XR 8mg tablet once daily, orally up to 52 weeks. If a participant and caregiver chose to extend treatment beyond the first 52 weeks, following re-consent, participants were allowed to continue the treatment and attended visits at the following time points every year: 12, 24, 36 and 52 weeks.
Period: Overall Study
Arm/Group | RSG XR 8 mg
Started | 331
Completed | 26
Not Completed | 305
Not completed — Adverse Event | 28
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 11
Not completed — Withdrawal by Subject | 30
Not completed — Still in study at termination | 206
Not completed — Missing | 2
Not completed — Prolonged QT Interval Electrocardiogram | 12
Not completed — Investigators opinion | 1
Not completed — Lack of curative effect | 1
Not completed — Unethical stop of enrollment | 2
Not completed — Caregiver's decision to withdraw | 1
Not completed — Out of Electrocardiogram criteria | 1
Not completed — Exclusion criteria | 1
Not completed — Prohibited medicine | 1

BASELINE CHARACTERISTICS:
Groups:
- RSG XR 8 mg: Participants received RSG XR 4mg tablet once daily, orally for the first 4 weeks of the study followed by RSG XR 8mg tablet once daily, orally up to 52 weeks. If a participant and caregiver chose to extend treatment beyond the first 52 weeks, following re-consent, participants were allowed to continue the treatment and attended visits at the following time points every year: 12, 24, 36 and 52 weeks.
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 85
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 242
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Severity of AEs
Description: AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The drug related-AEs of special interest (AESI) was reported. The severity of the AESI was categorized as mild, moderate and severe. Number of participants with AEs were reported for treatment duration of the study.
Time Frame: Up to Week 82
Population: All subject population was comprised of all participants who took at least one dose of open-label study medication.
Measure: Count of Participants; unit: Participants
Groups:
- RSG XR 8mg: Participants received RSG XR 4mg tablet once daily, orally for the first 4 weeks of the study followed by RSG XR 8mg tablet once daily, orally up to 52 weeks. If a participant and caregiver chose to extend treatment beyond the first 52 weeks, following re-consent, participants were allowed to continue the treatment and attended visits at the following time points every year: 12, 24, 36 and 52 weeks.
Arm/Group | RSG XR 8mg
Number analyzed (Participants) | 331
Participants
  Any AEs | 125
  Total Drug-Related AESI | 46
  Mild AESI | 31
  Moderate AESI | 13
  Severe AESI | 2

2. Secondary Outcome: Number of Participants With Serious AEs and Deaths
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose results in death, life-threatening condition, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, or a congenital anomaly or birth defect. The SAEs and deaths are reported from Visit 1 (W0) till end of the follow-up period (W110)
Time Frame: Up to Week 82
Population: All subject population
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Participants
  Any SAE | 8
  Death | 3

3. Secondary Outcome: Percentage of Participants With AEs of Edema
Description: Edema was considered as adverse event of special interest (AESI). The process for AESI selection was based on RSG's pharmacologic class and relevant AEs potentially associated with RSG. Percentage of participants reported with edema as AESI were reported.
Time Frame: Up to 82 Weeks
Population: All subject population
Measure: Number; unit: Percentage of participants
Groups:
- RSG XR 8 mg: Participants received RSG XR 4 mg tablet orally once daily for first 4 weeks (W 0 to W 4) of treatment followed by RSG XR 8 mg tablet orally once daily from W 5 to W 104.
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Percentage of participants | 13

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP of participant were recorded in sitting posture as vital sign at each visit. The blood pressure (BP) values were identified as of potential clinical concern if the vales were out of the reference range (for SBP, 90 to 140 mmHg and DBP, 50 to 90 mmHg) or meet a change from Baseline criterion. The change from Baseline criterion for SBP, was increase from Baseline (high) if increased by more than or equal to (>=) 40 mmHg from Baseline; decrease from Baseline (low) if decreased by >= 30 mmHg from Baseline. For DBP, increase form Baseline (high) if increased by >= 30 mmHg from Baseline; decrease from Baseline (low) if decreased by >= 20 mmHg from Baseline. The Baseline assessments were referred to assessments at Visit 1 (W 0). Change from Baseline was measured as the blood pressure value recorded at specified visit minus the Baseline value.
Time Frame: Baseline (Visit 1, W0), W4, W8, W12, W16, W24, W36, W52, W64 and Follow-up (W82)
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
millimeter of mercury (mmHg)
  SBP, W4: number analyzed (Participants) | 318
  SBP, W4 | -0.2 (11.61)
  SBP, W8: number analyzed (Participants) | 294
  SBP, W8 | -1.1 (11.83)
  SBP, W12: number analyzed (Participants) | 281
  SBP, W12 | -0.7 (13.80)
  SBP, W16: number analyzed (Participants) | 271
  SBP, W16 | -1.3 (13.66)
  SBP, W24: number analyzed (Participants) | 231
  SBP, W24 | -1.2 (13.30)
  SBP, W36: number analyzed (Participants) | 134
  SBP, W36 | -3.0 (15.37)
  SBP, W52: number analyzed (Participants) | 37
  SBP, W52 | 0.3 (12.85)
  SBP, Year 2 W12: number analyzed (Participants) | 10
  SBP, Year 2 W12 | -0.1 (16.93)
  SBP, Follow-up: number analyzed (Participants) | 280
  SBP, Follow-up | -0.5 (12.32)
  DBP, W4: number analyzed (Participants) | 318
  DBP, W4 | -0.8 (7.59)
  DBP, W8: number analyzed (Participants) | 294
  DBP, W8 | -2.1 (8.52)
  DBP, W12: number analyzed (Participants) | 281
  DBP, W12 | -2.0 (8.74)
  DBP, W16: number analyzed (Participants) | 271
  DBP, W16 | -2.2 (9.00)
  DBP, W24: number analyzed (Participants) | 231
  DBP, W24 | -2.1 (8.53)
  DBP, W36: number analyzed (Participants) | 134
  DBP, W36 | -3.0 (9.11)
  DBP, W52: number analyzed (Participants) | 37
  DBP, W52 | -1.4 (8.26)
  DBP, Year 2 W12: number analyzed (Participants) | 10
  DBP, Year 2 W12 | 2.8 (9.86)
  DBP, Follow-up: number analyzed (Participants) | 280
  DBP, Follow-up | -0.9 (9.04)

5. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: HR of participants was recorded as vital sign at each visit. The HR values were identified as of potential clinical concern if the vales were out of the reference range 50 to 100 beats per minute (BPM) or meet a change from Baseline criterion. The change from Baseline criterion was as, increase in HR (high) from Baseline if HR was increased by >= 30 bpm or decrease in HR (Low) from Baseline if HR was decreased by >= 30 bpm from Baseline. The Baseline assessments were referred to assessments at Visit 1 (W 0). Change from Baseline was measured as the HR at specified visit minus the Baseline value.
Time Frame: Baseline (Visit 1, W0), W4, W8, W12, W16, W24, W36, W52, W64 and Follow-up (W82)
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | RSG XR 8mg
Number analyzed (Participants) | 331
BPM
  HR, W4: number analyzed (Participants) | 318
  HR, W4 | 1.1 (7.19)
  HR, W8: number analyzed (Participants) | 294
  HR, W8 | 1.8 (7.44)
  HR, W12: number analyzed (Participants) | 281
  HR, W12 | 2.2 (8.70)
  HR, W16: number analyzed (Participants) | 271
  HR, W16 | 1.2 (7.89)
  HR, W24: number analyzed (Participants) | 231
  HR, W24 | 1.0 (7.87)
  HR, W36: number analyzed (Participants) | 134
  HR, W36 | 1.7 (7.60)
  HR, W52: number analyzed (Participants) | 37
  HR, W52 | -0.8 (8.87)
  HR, Year 2 W12: number analyzed (Participants) | 10
  HR, Year 2 W12 | 2.9 (10.64)
  HR, Follow-up: number analyzed (Participants) | 280
  HR, Follow-up | 1.6 (8.17)

6. Secondary Outcome: Number of Participants With Abnormal SBP and DBP at Any Time During Treatment Period
Description: as for outcome 4
Time Frame: Up to 82 weeks
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Participants
  SBP, >140 or <90, | 84
  SBP, Increase from Baseline >=40, | 8
  SBP, Decrease from Baseline >=30, | 22
  DBP, >90 or <50, | 23
  DBP, Increase from Baseline >=30, | 2
  DBP, Decrease from Baseline >=20, | 31

7. Secondary Outcome: Number of Participants With Abnormal HR at Any Time During Treatment Period
Description: HR of participants was recorded as vital sign at each visit. The HR values were identified as of potential clinical concern if the vales were out of the reference range 50 to 100 beats per minute (BPM) or meet a change from Baseline criterion. The change from Baseline criterion was as, increase in HR (high) from Baseline if HR was increased by >= 30 bpm or decrease in HR (Low) from Baseline if HR was decreased by >= 30 bpm from Baseline. The Baseline assessments were referred to assessments at Visit 1 (W 0). Change from Baseline was measured as the HR at specified visit minus the Baseline value. Number of participants with abnormal HR at any time during treatment period were reported.
Time Frame: Up to 82 weeks
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 319
Participants
  HR, >100 or <50 | 3
  HR, Increase from baseline >=30 | 2

8. Secondary Outcome: Change From Baseline in Body Weight (BW)
Description: BW of participants were recorded as vital sign at each visit. The BW were identified as of potential clinical concern if the vales were increased or decreased from Baseline by >=7%. The Baseline assessments were referred to assessments at Visit 1 (W0). Change from Baseline was measured as the BW at specified visit minus the Baseline value.
Time Frame: Baseline (Visit 1, W0), W4, W8, W12, W16, W24, W36, W52, W64 and Follow-up (W82)
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Kilograms (kg)
  BW, W4: number analyzed (Participants) | 318
  BW, W4 | 0.2 (1.57)
  BW, W8: number analyzed (Participants) | 293
  BW, W8 | 0.4 (2.42)
  BW, W12: number analyzed (Participants) | 281
  BW, W12 | 0.5 (2.06)
  BW, W16: number analyzed (Participants) | 271
  BW, W16 | 0.5 (2.59)
  BW, W24: number analyzed (Participants) | 231
  BW, W24 | 0.6 (2.80)
  BW, W36: number analyzed (Participants) | 134
  BW, W36 | 0.5 (3.60)
  BW, W52: number analyzed (Participants) | 37
  BW, W52 | -0.0 (3.75)
  BW, Year 2 W12: number analyzed (Participants) | 10
  BW, Year 2 W12 | 0.5 (3.92)
  BW, Follow-up: number analyzed (Participants) | 280
  BW, Follow-up | 0.5 (3.04)

9. Secondary Outcome: Number of Participants With Abnormal BW at Any Time During Treatment Period
Description: BW of participants were recorded as vital sign at each visit. The BW were identified as of potential clinical concern if the vales were increased or decreased from Baseline by >=7%. The Baseline assessments were referred to assessments at Visit 1 (W0). Change from Baseline in BW was measured as the BW value at specified visit minus the Baseline BW value. Number of participants with abnormal BW at any time during treatment period were reported.
Time Frame: Baseline (Visit 1, W0) to W 52
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 318
Participants
  Increase from Baseline >=7% | 30
  Decrease from Baseline >=7% | 16

10. Secondary Outcome: Change From Baseline in Non-fasting Measures of Lipid Metabolism Including Total Cholesterol, High Density Lipoprotein, Low Density Lipoprotein and Triglycerides at Indicated Timepoints.
Description: Non-fasting measures of lipid metabolism including cholesterol (TC), high density lipoprotein (HDL), low density lipoprotein (LDL), triglycerides (TG) were measured at Baseline (W0), W4, W16, W36, W52, Year 2 W24 and Follow-up. The Baseline assessments were referred to assessments at Visit 1 (W0). Change from Baseline was calculated as the value at the indicated visit minus the Baseline value.
Time Frame: Baseline (Visit 1, W0), W4, W16, W36, W52, W76, and W82
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per litre
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Millimoles per litre
  TC, W4: number analyzed (Participants) | 288
  TC, W4 | 0.106 (0.7341)
  TC, W16: number analyzed (Participants) | 254
  TC, W16 | 0.200 (0.9713)
  TC, W36: number analyzed (Participants) | 142
  TC, W36 | 0.140 (1.0659)
  TC, W52: number analyzed (Participants) | 35
  TC, W52 | 0.333 (1.2454)
  TC, Year 2 W24: number analyzed (Participants) | 8
  TC, Year 2 W24 | 1.163 (0.6604)
  TC, Follow-up: number analyzed (Participants) | 134
  TC, Follow-up | 0.069 (0.9649)
  HDL, W4: number analyzed (Participants) | 288
  HDL, W4 | -0.035 (0.2217)
  HDL, W16: number analyzed (Participants) | 254
  HDL, W16 | -0.030 (0.2597)
  HDL, W36: number analyzed (Participants) | 142
  HDL, W36 | -0.069 (0.2711)
  HDL, W52: number analyzed (Participants) | 35
  HDL, W52 | -0.020 (0.3420)
  HDL, Year 2 W24: number analyzed (Participants) | 8
  HDL, Year 2 W24 | -0.150 (0.4104)
  HDL, Follow-up: number analyzed (Participants) | 134
  HDL, Follow-up | -0.057 (0.2325)
  LDL, W4: number analyzed (Participants) | 281
  LDL, W4 | 0.088 (0.6689)
  LDL, W16: number analyzed (Participants) | 248
  LDL, W16 | 0.211 (0.9151)
  LDL, W36: number analyzed (Participants) | 140
  LDL, W36 | 0.163 (0.9484)
  LDL, W52: number analyzed (Participants) | 34
  LDL, W52 | 0.385 (1.0346)
  LDL, Year 2 W24: number analyzed (Participants) | 8
  LDL, Year 2 W24 | 1.051 (0.5836)
  LDL, Follow-up: number analyzed (Participants) | 132
  LDL, Follow-up | 0.133 (0.8985)
  TG, W4: number analyzed (Participants) | 288
  TG, W4 | 0.084 (0.6918)
  TG, W16: number analyzed (Participants) | 254
  TG, W16 | 0.027 (0.8355)
  TG, W36: number analyzed (Participants) | 142
  TG, W36 | 0.050 (0.8774)
  TG, W52: number analyzed (Participants) | 35
  TG, W52 | -0.179 (1.0565)
  TG, Year 2 W24: number analyzed (Participants) | 8
  TG, Year 2 W24 | 0.573 (0.8992)
  TG, Follow-up: number analyzed (Participants) | 134
  TG, Follow-up | -0.062 (0.7616)

11. Secondary Outcome: Number of Participants With Hematological Parameters of Potential Clinical Concern
Description: The hematological parameters including eosinophils, lymphocytes, monocytes, platelet count, Segmented Neutrophils, total neutrophils, white blood cell (WBC), red blood cell (RBC) counts, hemoglobin, hematocrit count, mean corpuscle hemoglobin (MCH) and mean corpuscle volume (MCV) were analyzed as safety parameters. The number of participants with values outside the reference range (potential clinical concern ) at any time on treatment (ATOT) and follow-up period were reported. The treatment period was till W104 followed by 6 weeks of follow-up period till W110 of study.
Time Frame: Up to 82 weeks
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Participants
  Eosinophils, ATOT, High: number analyzed (Participants) | 308
  Eosinophils, ATOT, High | 1
  Hematocrit, ATOT, Low: number analyzed (Participants) | 308
  Hematocrit, ATOT, Low | 2
  Hematocrit, Follow-up, Low: number analyzed (Participants) | 139
  Hematocrit, Follow-up, Low | 1
  Hemoglobin, ATOT, High: number analyzed (Participants) | 308
  Hemoglobin, ATOT, High | 1
  Hemoglobin, ATOT, Low: number analyzed (Participants) | 308
  Hemoglobin, ATOT, Low | 20
  Hemoglobin, Follow-Up, Low: number analyzed (Participants) | 139
  Hemoglobin, Follow-Up, Low | 8
  Lymphocytes, ATOT, Low: number analyzed (Participants) | 308
  Lymphocytes, ATOT, Low | 5
  Lymphocytes, Follow-Up, Low: number analyzed (Participants) | 137
  Lymphocytes, Follow-Up, Low | 3
  MCH, ATOT, High: number analyzed (Participants) | 308
  MCH, ATOT, High | 1
  MCH, Follow-Up, High: number analyzed (Participants) | 139
  MCH, Follow-Up, High | 1
  MCV, ATOT, High: number analyzed (Participants) | 308
  MCV, ATOT, High | 1
  MCV, Follow-Up, High: number analyzed (Participants) | 139
  MCV, Follow-Up, High | 1
  Monocytes, ATOT, Low: number analyzed (Participants) | 308
  Monocytes, ATOT, Low | 17
  Monocytes, ATOT, High: number analyzed (Participants) | 137
  Monocytes, ATOT, High | 5
  Platelet count, ATOT, High: number analyzed (Participants) | 308
  Platelet count, ATOT, High | 1
  Platelet count, ATOT, Low: number analyzed (Participants) | 308
  Platelet count, ATOT, Low | 2
  Red Cell Distribution Width, ATOT, High: number analyzed (Participants) | 308
  Red Cell Distribution Width, ATOT, High | 30
  Red Cell Distribution Width,Follow-up, High: number analyzed (Participants) | 139
  Red Cell Distribution Width,Follow-up, High | 8
  Red Blood Cell count, ATOT, Low: number analyzed (Participants) | 308
  Red Blood Cell count, ATOT, Low | 4
  Red Blood Cell count, Follow-up, Low: number analyzed (Participants) | 139
  Red Blood Cell count, Follow-up, Low | 4
  Segmented Neutrophils, ATOT, High: number analyzed (Participants) | 308
  Segmented Neutrophils, ATOT, High | 1
  Segmented Neutrophils, ATOT, Low: number analyzed (Participants) | 308
  Segmented Neutrophils, ATOT, Low | 14
  Segmented Neutrophils, Follow-up, Low: number analyzed (Participants) | 137
  Segmented Neutrophils, Follow-up, Low | 2
  Total Neutrophils, ATOT, High: number analyzed (Participants) | 308
  Total Neutrophils, ATOT, High | 1
  Total Neutrophils, ATOT, Low: number analyzed (Participants) | 308
  Total Neutrophils, ATOT, Low | 14
  Total Neutrophils, Follow-Up, Low: number analyzed (Participants) | 137
  Total Neutrophils, Follow-Up, Low | 2
  WBC, ATOT, Low: number analyzed (Participants) | 308
  WBC, ATOT, Low | 9

12. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters of Potential Clinical Concern
Description: The clinical chemistry parameters including alanine amino transferase (ALT), aldolase, aspartate amino transferase (AST), blood urea nitrogen /creatinine (BUN/Creat) ratio, cholesterol (Chol), creatine kinase, creatinine, direct bilirubin, gamma glutamyl transferase (GGT), glucose, high density lipid (HDL), low density lipid (LDL), potassium, troponin 1, and urea were assessed as safety parameters. The number of participants with values outside the reference range (potential clinical concern ) at any time on treatment (ATOT) and follow-up period were reported. The treatment period was till W104 followed by 6 weeks of follow-up period till W110 of study.
Time Frame: Up to 82 weeks
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Participants
  ALT, ATOT, High: number analyzed (Participants) | 309
  ALT, ATOT, High | 1
  ALT, Follow-up, High: number analyzed (Participants) | 142
  ALT, Follow-up, High | 1
  Aldolase, ATOT, High: number analyzed (Participants) | 56
  Aldolase, ATOT, High | 3
  Aldolase, ATOT, Low: number analyzed (Participants) | 56
  Aldolase, ATOT, Low | 7
  Aldolase, Follow-up, Low: number analyzed (Participants) | 24
  Aldolase, Follow-up, Low | 3
  AST, ATOT, High: number analyzed (Participants) | 309
  AST, ATOT, High | 2
  AST, Follow-up, High: number analyzed (Participants) | 142
  AST, Follow-up, High | 1
  BUN/Creat ratio, ATOT, High: number analyzed (Participants) | 309
  BUN/Creat ratio, ATOT, High | 18
  BUN/Creat ratio, Follow-up, High: number analyzed (Participants) | 142
  BUN/Creat ratio, Follow-up, High | 1
  Chol, ATOT, High: number analyzed (Participants) | 309
  Chol, ATOT, High | 52
  Chol, Follow-up, High: number analyzed (Participants) | 142
  Chol, Follow-up, High | 13
  Creatine Kinase, ATOT, High: number analyzed (Participants) | 309
  Creatine Kinase, ATOT, High | 32
  Creatine Kinase, Follow-up, High: number analyzed (Participants) | 142
  Creatine Kinase, Follow-up, High | 7
  Creatinin, ATOT, High: number analyzed (Participants) | 309
  Creatinin, ATOT, High | 4
  Creatinin, Follow-up, High: number analyzed (Participants) | 142
  Creatinin, Follow-up, High | 5
  Direct Bilirubin, ATOT, High: number analyzed (Participants) | 309
  Direct Bilirubin, ATOT, High | 1
  GGT, ATOT, High: number analyzed (Participants) | 309
  GGT, ATOT, High | 308
  GGT, Follow-up, High: number analyzed (Participants) | 142
  GGT, Follow-up, High | 142
  Glucose, ATOT, High: number analyzed (Participants) | 309
  Glucose, ATOT, High | 19
  Glucose, ATOT, Low: number analyzed (Participants) | 309
  Glucose, ATOT, Low | 5
  Glucose, Follow-up, High: number analyzed (Participants) | 142
  Glucose, Follow-up, High | 8
  HDL, ATOT, Low: number analyzed (Participants) | 309
  HDL, ATOT, Low | 1
  LDL, ATOT, High: number analyzed (Participants) | 307
  LDL, ATOT, High | 135
  LDL, Follow-up, High: number analyzed (Participants) | 142
  LDL, Follow-up, High | 45
  Potassium, ATOT, High: number analyzed (Participants) | 309
  Potassium, ATOT, High | 4
  Potassium, ATOT, Low: number analyzed (Participants) | 309
  Potassium, ATOT, Low | 1
  Troponin I, ATOT, High: number analyzed (Participants) | 47
  Troponin I, ATOT, High | 2
  Urea, ATOT, High: number analyzed (Participants) | 309
  Urea, ATOT, High | 19
  Urea, Follow-up, High: number analyzed (Participants) | 142
  Urea, Follow-up, High | 7

13. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) Total Score as a Function of Apolipoprotein E (APOE) 4 Status at W24 and W52
Description: The 11-item ADAS-cog was used to assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores ranged from 0 to 70 with higher scores indicating greater dysfunction. Baseline was referred to Visit 1 (W0)assessments. Change from Baseline was calculated as value at scheduled time point minus Baseline value.
Time Frame: Baseline (Visit 1, W0), W24 and W52
Population: All subject population. All subject population was further stratified to 4 different cohorts based upon APOE 4 status as APOE 4 negative, APOE 4 positive, APOE 4 heterozygus and APOE 4 homozygus. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Score on scale
  All subject population, W24: number analyzed (Participants) | 243
  All subject population, W24 | 1.9 (5.23)
  All subject population, W52: number analyzed (Participants) | 58
  All subject population, W52 | 2.5 (5.69)
  APOE4, Neg, W24: number analyzed (Participants) | 115
  APOE4, Neg, W24 | 2.1 (5.29)
  APOE4, Neg, W52: number analyzed (Participants) | 32
  APOE4, Neg, W52 | 3.0 (5.40)
  APOEe4, Pos, W24: number analyzed (Participants) | 128
  APOEe4, Pos, W24 | 1.8 (5.19)
  APOEe4, Pos, W52: number analyzed (Participants) | 26
  APOEe4, Pos, W52 | 1.8 (6.07)

14. Secondary Outcome: Mean Clinician Interview-Based Impression of Change Plus Caregiver Input (CIBIC+) Score as a Function of APOE 4 Status
Description: The CIBIC+ score used for global functioning assessment. The CIBIC+ assessment comprised of a 7-point rating of severity. It was rated on a scale of 1 to 7 as 1: markedly improved, 2.: moderately improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: moderately worse and 7: markedly worse; The lower score indicated betterment in functioning and higher score means greater dysfunction. The scale was based on interviews with the participant and the caregiver and was completed by an independent rater.
Time Frame: Baseline (Visit 1, W0), W 24 and W 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Score on scale
  All subject population, W24: number analyzed (Participants) | 241
  All subject population, W24 | 4.3 (1.05)
  All subject population, W52: number analyzed (Participants) | 60
  All subject population, W52 | 4.5 (1.10)
  APOEe4, Neg, W24: number analyzed (Participants) | 113
  APOEe4, Neg, W24 | 4.3 (1.04)
  APOEe4, Neg, W52: number analyzed (Participants) | 33
  APOEe4, Neg, W52 | 4.7 (1.16)
  APOEe4, Pos, W24: number analyzed (Participants) | 128
  APOEe4, Pos, W24 | 4.3 (1.05)
  APOEe4, Pos, W52: number analyzed (Participants) | 27
  APOEe4, Pos, W52 | 4.3 (0.99)

15. Secondary Outcome: Change From Baseline in Mini Mental State Examination (MMSE) Total Score as a Function of APOE 4 Status at W24 and W52
Description: The MMSE consisted of 11 tests of orientation, memory (recent and immediate), concentration, language and praxis. Scores range from 0 to 30, with lower scores indicating greater cognitive impairment. The scale was completed by the investigator, based on the performance of the participant, and took approximately 5 to 10 minutes to administer. Change from parent Baseline in MMSE was analyzed using a mixed model for repeated measures (MMRM). Baseline was referred to Visit 1 (W0)assessments. Change from Baseline was calculated as value at scheduled time point minus Baseline value.
Time Frame: Baseline (Visit 1, W0), W 24 and W52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Score on scale
  All subject population, W24: number analyzed (Participants) | 203
  All subject population, W24 | -0.7 (2.65)
  All subject population, W52: number analyzed (Participants) | 19
  All subject population, W52 | -1.6 (2.85)
  APOEe4, Neg, W24: number analyzed (Participants) | 91
  APOEe4, Neg, W24 | -0.7 (2.70)
  APOEe4, Neg, W52: number analyzed (Participants) | 11
  APOEe4, Neg, W52 | -1.2 (3.37)
  APOEe4, Pos, W24 | -0.7 (2.63)
  APOEe4, Pos, W52: number analyzed (Participants) | 8
  APOEe4, Pos, W52 | -2.1 (2.03)

16. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia Scale (DAD) Total Score as a Function of APOEe 4 Status
Description: The DAD, assessed the ability of a participant to execute basic and instrumental activities of daily living (ADL) and leisure activities. The scale consists of 40 questions assessing basic and instrumental ADLs. This scale assesses a participant's ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item was scored as yes: 1, no: 0 and N/A: not applicable. Higher scores indicate less disability with a score of 100 indicating no disability and 0 indicating no functional ability. The percentage score was calculated as (DAD total score/total number of applicable items) multiplied by 100. The DAD was conducted as an interview with the caregiver and took approximately 20 minutes. Baseline was referred to Visit 1 (W0) assessments. Change from Baseline was calculated as value at scheduled time point minus Baseline value.
Time Frame: Baseline (Visit 1, W0), W24 and W52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Score on scale
  All subject population, W24: number analyzed (Participants) | 203
  All subject population, W24 | -3.2 (10.23)
  All subject population, W52: number analyzed (Participants) | 19
  All subject population, W52 | -5.2 (18.21)
  APOEe4, Neg, W24: number analyzed (Participants) | 91
  APOEe4, Neg, W24 | -4.5 (11.57)
  APOEe4, Neg, W52: number analyzed (Participants) | 11
  APOEe4, Neg, W52 | -6.2 (22.66)
  APOEe4, Pos, W24: number analyzed (Participants) | 112
  APOEe4, Pos, W24 | -2.2 (8.91)
  APOEe4, Pos, W52: number analyzed (Participants) | 8
  APOEe4, Pos, W52 | -3.8 (10.73)

17. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score as a Function of APOE 4 Status at W24 and W52
Description: The NPI assessed behavioural disturbances comprises 10 dimensions: delusions, hallucinations, dysphoria, apathy, euphoria, disinhibition, aggressiveness and agitation, irritability, anxiety and aberrant motor activity. The participant caregiver asked about behaviour in the participant. If "Yes", the informant then rates both the severity on a 3-point scale, 1: mild to 3: severe (total range: 0-36) and the frequency using a 4-point scale, 1: occasionally to 4: very frequently. The total domain score was frequency × severity. The distress was scored on 5-point scale, 0: no distress to 5 - very severe or extreme. A total NPI score was calculated by adding all domain scores together: NPI total score (from 0-144) and NPI distress score (from 0-60), with higher scores indicating more severe behavioral disturbance. Baseline was referred to Visit 1 (W0) assessments. Change from Baseline was calculated as value at scheduled time point minus Baseline value.
Time Frame: Baseline (Visit 1, W0), W24 and W52
Population: All subject population. All subject population was further stratified to 4 different cohorts based upon APOE 4 status as APOE 4 negative, APOE 4 positive, APOE 4 heterozygus and APOE 4 homozygus. Only those participants available at the indicated time points were analyzed (represented by n=X, X, X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Score on scale
  All subject population, W24: number analyzed (Participants) | 203
  All subject population, W24 | 1.1 (7.07)
  All subject population, W52: number analyzed (Participants) | 19
  All subject population, W52 | 2.1 (9.55)
  APOEe4, Neg, W24: number analyzed (Participants) | 91
  APOEe4, Neg, W24 | 1.9 (8.24)
  APOEe4, Neg, W52: number analyzed (Participants) | 11
  APOEe4, Neg, W52 | 1.5 (9.41)
  APOEe4, Pos, W24: number analyzed (Participants) | 112
  APOEe4, Pos, W24 | 0.4 (5.91)
  APOEe4, Pos, W52: number analyzed (Participants) | 8
  APOEe4, Pos, W52 | 2.8 (10.35)

18. Secondary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: HbA1c was evaluated as safety parameter in this study. The values of change from Baseline was presented. The Baseline assessments were referred to assessments at Visit 1 (W0). Change from Baseline was measured as the BW at specified visit minus the Baseline value.
Time Frame: Baseline (Vsit 1 W0), W12, W24, W36, W52, W76 and Follow-up (W82)
Population: All subject population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | RSG XR 8 mg
Number analyzed (Participants) | 331
Percent HbA1c
  W12: number analyzed (Participants) | 61
  W12 | -0.02 (0.573)
  W24: number analyzed (Participants) | 65
  W24 | 0.08 (0.512)
  W36: number analyzed (Participants) | 59
  W36 | 0.03 (0.417)
  W52: number analyzed (Participants) | 29
  W52 | 0.09 (0.377)
  W76: number analyzed (Participants) | 8
  W76 | 0.08 (0.369)
  Follow-up: number analyzed (Participants) | 95
  Follow-up | 0.07 (0.540)

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-SAEs were collected during the treatment period (up to 82 weeks)
Description: On-treatment SAEs and non-serious AEs were reported for the All subject population consisted of all participants who received at least one dose of study drug.
Arm/Group | RSG XR 8 mg
All-Cause Mortality (participants affected / at risk) | 3/331
Serious Adverse Events (participants affected / at risk) | 8/331
Other Adverse Events (participants affected / at risk) | 42/331
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSG XR 8 mg (N=331)
Atrioventricular block complete (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Facial palsy (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Atrial fibrillation (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Mental impairment (Nervous system disorders) | 1
Crush syndrome (Renal and urinary disorders) | 1
Circulatory collapse (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RSG XR 8 mg (N=331)
Oedema peripheral (General disorders) | 42 — General disorders and administration site conditions

LIMITATIONS AND CAVEATS:
The study was early terminated on 12 February 2009 because RSG XR as monotherapy in Alzheimer's disease failed to demonstrate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.